CLINICAL TRIAL: NCT05800548
Title: The Relationship Between Health Literacy and Family Planning Attitudes of Postpartum Women
Brief Title: Health Literacy of Postpartum Women and Family Planing
Status: Completed | Type: Observational
Sponsor: Osmaniye Korkut Ata University (Other)
Collaborators: Mersin University (Other)
Responsible Party: Principal Investigator, Derya Kaya Senol, Principal Investigator, Osmaniye Korkut Ata University
Other Study IDs: DKSenol
Record Dates: First submitted 2022-10-04; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Contraception; Health Attitude; Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- postpartum women: The sample of the research is; puerperant women who applied to the hospital for delivery within the research dates and gave birth in a healthy way, did not have any risk for the mother and the baby, had no communication barriers and met the research criteria.
  Interventions: Other: survey application

INTERVENTIONS:
Other: survey application — In data collection; Socio-demographic and obstetric characteristics of puerperant women, descriptive information form including questions about current birth, Postpartum Family Planning Attitude Scale The Health Literacy Scale was used.

SUMMARY:
This study was carried out as a cross-sectional-relationship searcher in order to determine the effect of evaluating the relationship between health literacy and family planning attitudes of postpartum women.

The population of the study consisted of puerperant women in the Postpartum Clinic of Osmaniye State Hospital between March 2022 and June 2022. The sample of the research is; puerperant women who applied to the hospital for delivery within the research dates and gave birth in a healthy way, did not have any risk for the mother and the baby, had no communication barriers and met the research criteria. The sample number of the study was calculated using the G*Power 3.1.9.4 program.

The puerperant women who met the inclusion criteria were included in the study with the method of improbable random sampling, and a total of 258 puerperant women were reached.

In data collection; Socio-demographic and obstetric characteristics of puerperant women, descriptive information form including questions about current birth, Postpartum Family Planning Attitude Scale The Health Literacy Scale was used. In the study, a very strong positive correlation was found between the women's total PAPTS score and SAS total score (p=0.000). In other words; As the health literacy levels of postpartum women increase, their family planning attitude levels also increase

DETAILED DESCRIPTION:
Prior to the collection of research data, written permission was obtained from the institution where the research was conducted. On the first page of the survey, which was prepared by the researchers based on the literature review, puerperal women were informed about the study and their written consent was received. Data collection instruments were applied through face-to-face interviews to puerperal women in their own rooms in the clinic, at an appropriate time period for the infants and themselves. The application took approximately 10 to 15 minutes for each participant.

Data collection instruments The Mother Introductory Information Form (MIIF), consisting of questions about sociodemographic and obstetric characteristics, and the last delivery of puerperal mothers, the Postpartum Family Planning Attitude Scale (PFPAS), and the Health Literacy Scale (HLS) were used for data collection.

The MIIF was prepared by the researchers in accordance with the literature (Berkman et al., 2011; Yee and Simon 2014., Maricic et al., 2020). The form consists of a total of 17 questions aim to determine the sociodemographic and reproductive characteristics of the mothers.

The PFPAS, developed by Varol in 2019, includes 27 items scored on a 5-Likert type scale. 16 of the items consist of positive statements, while 11 items consist of negative statements. In order to ensure consistency in the evaluation, negative statements are reverse coded. The scale items are scored ranging from 1 to 5. Positive statements are scored as 1=Strongly disagree, 2= Disagree, 3= Neutral, 4= Agree, and 5= Strongly agree, while negative statements are scored as 5=Strongly disagree, 4=Disagree, 3= Neutral, 2= Agree, and 1= Strongly agree. The scale consists of a total of six subscales as "Perceived Risk" (Items 1, 2, 3), "Perceived Seriousness" (Items 4, 5, 6), "Perceived Benefits" (Items 7, 8, 9, 10), "Perceived Obstacles" (Items 11, 12, 13, 14, 15, 16, 17, 18), "Taking Action" (Items 19, 20, 21, 22, 23), and "Self-Efficacy" (Items 24, 25, 26, 27). The lowest score to be obtained from the scale is 27, while the highest score is 135. Higher scores indicate higher level of health belief in terms of perceived risk, perceived seriousness, perceived obstacles, perceived benefits, taking action and self-efficacy, which is also associated with a positive attitude toward FP. The Cronbach's alpha coefficient of the original scale is 0.878 (Varol, 2019). The Cronbach's alpha coefficient calculated in the current study is 0.932.

The HLS, developed by Sorensen et al., (2013), consists of 47 items and two dimensions. It was then simplified by Toçi et al., (2013), and its validity and reliability were tested. The validity and reliability study of the Turkish version, consisting of 25 items, was conducted by Aras and Temel in 2017. The scale includes four subscales as Access to Information, Understanding Information, Appraisal / Assessment, and Application / Use. The items are scored on a 5-point range as "5: No difficulty, 4: A little bit of difficulty, 3: Moderate difficulty, 2: Quite a bit of difficulty, 1: Extreme difficulty or unable to perform activity". All items include positive statements. The lowest possible score to be obtained from the scale is 25, and the highest possible score is 125. Higher scores indicate higher level of HL, while lower scores indicate inadequate, problematic and weak level of HL. The Cronbach's alpha value of the original scale is 0.92, while it ranges between 0.62 and 0.79 in the subscales (Aras & Temel, 2017). It has been found 0.920 in the current study.

ELIGIBILITY:
Inclusion Criteria:

* Puerperant women who applied to the hospital for delivery within the research dates and gave birth in a healthy way,
* Did not have any risk for the mother and the baby,
* Had no communication barriers

Exclusion Criteria:

* Those who have any health problems of the mother and the baby,
* İlliterate,
* Communication barrier

Ages: 19 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — puerperant women
Study Population: The puerperant women who met the inclusion criteria were included in the study with the method of improbable random sampling, and a total of 258 puerperant women were reached.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Postpartum Family Planning Attitude Scale | 4 month
  In the study, a very strong positive correlation was found between the women's total Postpartum Family Planning Attitude Scale The Health Literacy Scale total score (p=0.000). In other words; As the health literacy levels of postpartum women increase, their family planning attitude levels also increase

CONTACTS AND LOCATIONS:
Locations (1):
- Derya Kaya Şenol, Osmaniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No